CLINICAL TRIAL: NCT04962672
Title: Anesthesia Induced Brain Cancer Survival (ABC Survival): A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 21-5527.0
Record Dates: First submitted 2021-05-19; First posted 2021-07-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia; Brain Cancer; Survival
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Experimental): 20 patients scheduled for the elective craniotomy for suspected high-grade gliomas resection will be enrolled and further randomized to receive total intravenous anesthesia (propofol group). Standard fasting and monitoring guidelines will be instituted. All patients will be induced and intubated after administration of intravenous boluses of fentanyl, propofol and rocuronium. For the maintenance phase of anesthesia, patients in the propofol group will receive continuous infusions of propofol and remifentanil. No patients will receive nitrous oxide.
  Interventions: Drug: Propofol group
- Sevoflurane group (Active Comparator): 20 patients scheduled for the elective craniotomy for suspected high-grade gliomas resection will be enrolled and further randomized to receive Volatile (sevoflurane group) agent for the maintenance phase of anesthesia. Standard fasting and monitoring guidelines will be instituted. All patients will be induced and intubated after administration of intravenous boluses of fentanyl, propofol and rocuronium. For the maintenance phase of anesthesia, patients in the volatile inhalational anesthesia group will received a volatile inhalational agent (sevoflurane) and remifentanil infusion. No patients will receive nitrous oxide.
  Interventions: Drug: Sevoflurane group

INTERVENTIONS:
Drug: Propofol group — 20 patients scheduled for the elective craniotomy for suspected high-grade gliomas resection will be enrolled and further randomized to receive total intravenous anesthesia (propofol group). Standard fasting and monitoring guidelines will be instituted. All patients will be induced and intubated after administration of intravenous boluses of fentanyl, propofol and rocuronium. For the maintenance phase of anesthesia, patients in the propofol group will receive continuous infusions of propofol and remifentanil. No patients will receive nitrous oxide. Anesthesia will be titrated to keep depth of anesthesia between 35- 55. All patients will be maintained on oxygen in air mixture (40%) and titrate the End Tidal Carbon Dioxide (ETCO2) concentration between 25-30 mm Hg.
  Other Names: Total intravenous anesthesia
  Arms: Propofol group
Drug: Sevoflurane group — 20 patients scheduled for the elective craniotomy for suspected high-grade gliomas resection will be enrolled and further randomized to receive Volatile (sevoflurane group) agent for the maintenance phase of anesthesia. Standard fasting and monitoring guidelines will be instituted. All patients will be induced and intubated after administration of intravenous boluses of fentanyl, propofol and rocuronium. For the maintenance phase of anesthesia, patients in the volatile inhalational anesthesia group received a volatile inhalational agent (sevoflurane) and remifentanil infusion. No patients will receive nitrous oxide. Anesthesia will be titrated to keep depth of anesthesia between 35- 55. All patients will be maintained on oxygen in air mixture (40%) and titrate the End Tidal Carbon Dioxide (ETCO2) concentration between 25-30 mm Hg.
  Other Names: Volatile anesthesia
  Arms: Sevoflurane group

SUMMARY:
Cancer is a leading cause of death worldwide. It is estimated that approximately 55,000 Canadians are surviving with brain tumors. It is projected that around 3000 persons will be diagnosed with brain and spinal cord tumors, and approximately 75 percent patients will not survive. Out of all brain cancers, high-grade gliomas [Glioblastoma Multiforme (GBM)] impose highest morbidity and mortality. Therefore, it is important to explore ways in which Investigators can improve and prolong the lives of patients suffering from brain cancers, particularly high-grade glioma, which is the most common and aggressive primary brain tumor.

So far the Investigators know that the surgery, chemotherapy and radiotherapy are the three corner stones management options for these patients, and majority of the research have been conducted on these three major domains. Therefore, it is imperative to explore the other variables those may impact survival characteristics. One of the integral variables of the brain cancer surgery is anesthesia. Interestingly, the role of anesthetics was explored in some other non-brain solid organ tumor surgeries. It is observed that out of the two main types of anesthesia [one is through intravenous (propofol) and other one is gaseous (sevoflurane)], intravenous based anesthesia maintenance regime may delay the cancer progression and prolong the recurrence free period. In addition, two very large retrospective studies with approximately 11,000 and 18,000 patients respectively, showed that as compared to gaseous (volatile anesthetics) based, intravenous (propofol) based anesthesia conferred some protection against cancer progression and was also associated with lesser overall mortality. The exact nature of these protective mechanisms is not known but in animal and other laboratory-based experiments, propofol seems to inhibit cancer formation steps, delays inflammation and provide protection from cancer cell growth. This is a feasibility study for knowing various aspects of workflow; recruitment characteristics of participants and various obstacles in implying anesthesia based protocols so that the Investigators can conduct a well-designed multicenter international randomized study.

DETAILED DESCRIPTION:
In Canada, cancer is the most common cause of death. Among solid organ cancers, brain tumors, depending upon type and grading, impose significant morbidity and mortality. In addition, cancer progression and recurrence is one of the most common complications in management of high-grade gliomas and among all, Glioblastoma Multiforme (GBM) is the most common and aggressive primary brain cancer. Many factors have been demonstrated to affect glioma progression . Some of the most consistently sited variables are age, grade of tumor, tumor size and location, molecular diagnosis, extent of resection, and chemotherapy and radiotherapy.

On the other hand, though, anesthesia remains an integral part of glioma surgeries, and two types of anesthetics (total intravenous agent, such as, propofol and volatile, such as sevoflurane) are commonly used during maintenance phase of general anesthesia (GA) across over all world; their effects on brain cancer progression are not yet investigated extensively. Recent studies have highlighted that there could be an association of anesthesia with cancer progression in other solid organs. Very few researches have been published demonstrating the relationship between type of anesthetic and glioma progression. One study found that exposure of glioblastoma stem cells to volatile agent (isoflurane) increased their migration capacity in vitro and increased their migration distance in vivo in animals. A second study found that exposure of glioma stem cells to sevoflurane increased tumor cell proliferation as well as tumor markers, most notably hypoxia-inducible factors (HIF), which are associated with cancer growth. Finally, a retrospective cohort study published in 2019 compared the progression free survival (PFS) of patients who underwent high-grade glioma surgery using two different types of anesthetics. They found that, for patients with low KPS, anesthesia maintenance with propofol yielded a longer PFS compared to sevoflurane (15). With this background, it seems propofol based anesthesia may limit the progression of brain cancer progression and therefore, the purpose is to evaluate type of anesthetics (propofol versus sevoflurane) as a factor responsible for glioma progression and survival characteristics. As the Investigators are planning for a future phase III study, it is imperative to understand thoroughly the details regarding feasibility, workflow, enrollment and drop out characteristics, reasons of deviation and adherence rates to anesthesia protocols and problems in follow ups. Therefore, this feasibility study is a path to a well-designed larger multicenter randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting between Jul 1, 2022 and Dec 28, 2023 for elective procedure
2. Males or females of >18 years
3. Patient will be undergoing primary craniotomy (with general anesthesia) for suspected high-grade primary glial brain tumor (WHO grade III and IV)

Exclusion Criteria:

1. Patients of pediatric age group and pregnant patients
2. Patients previously diagnosed with severe adrenal dysfunction (over activity or insufficiency)
3. Suspected low grade (grade I, II), glioma, tumors involving brainstem and optic tract, and as well as non-glial tumors (i.e. suspected brain metastasis)
4. Awake craniotomies
5. Any conditions that preclude postoperative MRI
6. Motor evoked potential monitoring or any other intraoperative condition that renders choice of anesthetics affected.
7. Recurrent GBM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 6 months
  Feasibility outcomes: successful recruitment of trial participants
retention rate | 6 months
  Feasibility outcomes: successful retention of trial participants
rate of protocol adherence | 6 months
  Feasibility outcomes: successful intervention fidelity, identification of barriers to implementation of the intervention, and the feasibility of collecting outcome assessment data.

SECONDARY OUTCOMES:
Overall survival | 6 months
  The following details will be monitored
  * date of detection of first progression,
  * after surgery radiotherapy (start day after surgery, dose, fractions),
  * after surgery chemotherapy (start date after surgery, number of cycles),
  * date of the last follow-up
Progression free survival | 6 months
  * date of detection of first progression,
  * after surgery radiotherapy (start day after surgery, dose, fractions),
  * after surgery chemotherapy (start date after surgery, number of cycles),
  * date of the last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Tumul Chowdhury, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital/UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No